CLINICAL TRIAL: NCT06389565
Title: Change My Story: Pilot Randomized Clinical Trial of Change My Story Among Young Persons Living With HIV and Depression
Brief Title: Change My Story Task Shifted Mental Health Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Ibadan (Other)
Responsible Party: Principal Investigator, Aimalohi Ahonkhai, Associate Physician in Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024p000857
Record Dates: First submitted 2024-04-09; First posted 2024-04-29 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Hiv; Depression; Psychological Distress
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PST alone (Active Comparator): Patients randomized to PST alone will receive PST delivered using a stepped-care approach. Subsequent care will be determined based on participant PHQ-9 score at the week 6 evaluation. All participants who do not achieve remission (PHQ-9 <12) after completion of the additional six-week therapy sessions, will be required to have a referral to either the general MD or psychiatrist at the clinic to determine need for pharmacologic treatment or additional intervention based on local clinical practice guidelines. During each PST session, the HIV counselor will ask the participant structured questions to identify those at risk of suicide, or with adverse reactions to prescribed antidepressants. Participants who indicate suicidality (plan/attempt) during PST sessions, or ongoing refractory disease (at reassessment points) will require immediate consultation by the psychiatry clinic.
  Interventions: Behavioral: Problem Solving Therapy
- PST with Change My Story (Experimental): In addition to all activities described in the PST alone arm, at enrollment, participants in the arm with Change My Story, will download the game onto their phones, receive instructions about the game and receive recommendations on how to play the game (at least one narrative for one of the three characters) each week within 48 hours of the PST session. Participants will be encouraged to set a weekly reminder alarm for their game play session. Participants will have an opportunity to explore the game at will according to these loose parameters prior to the first PST session.
  Interventions: Behavioral: Problem Solving Therapy; Other: Change My Story

INTERVENTIONS:
Behavioral: Problem Solving Therapy — Problem solving therapy (PST) is a cognitive-behavioral therapy (CBT)-based intervention that uses seven basic steps to teach problem solving orientation and skills to equip individuals to manage the impact of stressful life events on their mental health.
Other: Change My Story — Change My Story is a narrative game with a choose-your-own-adventure format in which players navigate emotionally difficult experiences along with the character(s) and interact with the virtual environment to choose a narrative path toward the story's conclusion. It will used to address important obstacles in the mental health treatment gap for Y-PLWH.
  Arms: PST with Change My Story

SUMMARY:
Psychological distress and depression are common among young people living with HIV (Y-PLWH) and negatively impact medication adherence and disease control. In low- and middle-income countries, this problem is compounded by the lack of trained mental health professionals on the provider side and the requirement of frequent clinic-based visits imposing greater cost, inconvenience, and stigma for patients. Change My Story, is a theory-grounded, interactive narrative game designed to address the key drivers of depression and psychological distress among Y-PLWH in Nigeria. This pilot hybrid implementation-effectiveness randomized controlled trial (RCT) will compare Change My Story combined with PST to PST alone among 80 Y-PLWH with depression or psychological distress.

DETAILED DESCRIPTION:
Young people living with HIV (Y-PLWH) have poor adherence to antiretroviral therapy and engagement in HIV care, making HIV the leading cause of death for African adolescents. Depression and psychological distress are much more common among Y-PLWH than in the general population, and are associated with significantly worse adherence to care and treatment when compared to Y-PLWH without these co-morbid conditions. Thus, untreated depression and severe psychological distress are important contributors to poor HIV outcomes in this population. Nigeria is home to the 4th largest HIV population globally and 10% of Y-PLWH, but mental health screening is not routinely conducted in this setting, and less than 10% of those diagnosed have access to evidence-based care. Despite this treatment gap, few interventions have targeted the mental health needs of Y-PLWH in Africa. The World Health Organization recommends that caregivers of Y-PLWH adopt youth-friendly strategies and incorporate psychosocial services to meet their needs, and that task shifting to non-specialized health workers be used to overcome the dearth of trained professionals in low and middle-income countries. Task-shifted problem Solving Therapy (PST) has been effectively used to treat both depression and psychological distress using a task-shifted approach. However, PST is an intensive strategy (typically 6-15 weekly sessions) often delivered in-person and poor completion rates are associated with less effectiveness -- a concern further magnified during the current COVID-19 climate. Mobile health technologies may be uniquely suited to surmount some of the obstacles for effective A theory-grounded game, Change My Story, has been developed which allows players navigate difficult experiences based on drivers of psychological distress and interact with a virtual environment this research aims to 1) conduct a hybrid implementation-effectiveness pilot RCT for 80 Y-PLWH with depression or psychological distress, and compare feasibility, acceptability, engagement, satisfaction and preliminary effectiveness among individuals receiving PST alone or PST with Change My Story, and 2) use the Consolidated Framework for Implementation Research (CFIR) to assess factors influencing engagement, acceptability, and satisfaction along with facilitators and barriers to implementation delivery.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* age 16-24 years
* self-reported proficiency in reading and understanding English.
* PHQ9 score of 8-17 and impairment in functioning (consistent with clinical depression)

Exclusion Criteria:

* pregnant or nursing
* in care and on ART for <6 months
* history of- or positive assessment for- bipolar or psychotic disorder.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Engagement | 3 months
  The percentage of recommended problem solving therapy sessions attended.
Patient Satisfaction with Interventionn | 3 months
  Based on an adapted version of the client satisfaction questionnaire (CSQ-8). Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Feasibility 1 | 3 months
  Weiner's feasibility of an intervention (FIM). Scales can be created for each measure by averaging responses. Scale values range from 1 to 5.
Feasibility 2 | 3 months
  Proportion of consented patients enrolled
Feasibility 3 | 3 months
  Proportion of game play sessions interrupted by technical problems
Feasibility 4 | 3 months
  Proportion of users requiring mobile phone (at baseline) or requiring a replacement phone (due to loss or theft)
Feasibility 5 | Baseline
  Proportion of users requiring mobile phone
Feasibility 6 | 3 months
  Proportion of users requiring mobile phone replacement due to loss or theft
Feasibility 7 | 3 months
  Proportion in need for additional data bundles
Acceptability 1 | Once
  Weiner's acceptability of an intervention. Scales can be created for each measure by averaging responses. Scale values range from 1 to 5.
Acceptability 2 | up to 3 months
  Number of minutes of total game play per month
Acceptability 3 | up to 3 months
  Number of days of total game play per month
Acceptability 4 | 3 months
  Percentage of recommended game play minutes completed
Acceptability 5 | 3 months
  Proportion of narratives completed assessed from aggregated game play metrics

SECONDARY OUTCOMES:
Remission of depression. | 3 and 6 months
  Patient health questionnaire-9. For this research, a PHQ-9 score < 6 will be considered in remission.
Remission of psychological distress. | 3 and 6 months
  Self reporting questionnaire-20. For this research, a SRQ-20 < 5 will be considered in remission.
ART adherence | 3 and 6 months
  Based on % pharmacy refill
Viral suppression | 3 and 6 months
  VL < 200 copies/mL

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ibadan, Ibadan, Oyo State, Nigeria

REFERENCES:
- [Derived] Eliazer C, Omotosho T, Kuti KM, Pierce LJ, Gray D, Audet CM, Awolude O, Gureje O, Oladeji B, Ahonkhai AA. A Mobile Game Intervention for Young Persons Living With HIV and Depression in Nigeria: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2025 Dec 3;14:e74199. doi: 10.2196/74199. PMID 41337738